CLINICAL TRIAL: NCT01154829
Title: Pan European Collaboration on Antipsychotic Naive Schizophrenia (PECANS): the Effects of D2 Antagonism on Candidate Endophenotypes
Brief Title: Pan European Collaboration on Antipsychotic Naive Schizophrenia (PECANS)
Acronym: PECANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); Rigshospitalet, Denmark (Other); Institute of Psychiatry, London (Other); UMC Utrecht (Other); Copenhagen Hospital Corporation (Other)
Responsible Party: Principal Investigator, Birte Glenthoj, professor, University of Copenhagen
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: H-D-2008-088
Record Dates: First submitted 2010-06-21; First posted 2010-07-01 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Schizophrenia
Keywords: dopamine; first episode; reward; cognition; MRI; fMRI; PPI; P300; P50 gating; endophenotypes
MeSH Terms: conditions — Schizophrenia | interventions — Amisulpride; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- first choice treatment (Active Comparator): Treatment with amisulpride
  Interventions: Drug: amisulpride
- second choice treatment (Active Comparator): treatment with aripiprazole
  Interventions: Drug: aripiprazole

INTERVENTIONS:
Drug: amisulpride — Individually dosed, according to symptoms, for a period of 6 weeks
  Other Names: Solian
  Arms: first choice treatment
Drug: aripiprazole — Individually dosed, according to symptoms, for a period of 6 weeks
  Other Names: abilify
  Arms: second choice treatment

SUMMARY:
The investigators want to relate disturbances in first-episode schizophrenic patients in (dopaminergic) D2 receptors, brain structure, brain function, and information processing to each other and to psychopathology. Additionally, the investigators want to examine the influence of D2 receptor blockade on these disturbances. The investigators expect disturbances in the dopaminergic system at baseline to correlate with specific structural and functional changes and with disruption in information processing as measured with psychophysiological and neurocognitive methods - and investigators expect D2 receptor blockade to reverse some of the functional and cognitive impairments.

DETAILED DESCRIPTION:
The study is designed as a 6 week case-control follow-up study of 70 AN FE pt. with SCZ and 70 controls matched with regard to age, gender, and parental socio-economic status. All subjects will be examined with a diagnostic interview (SCAN, Schedule for Clinical Assessment in Neuropsychiatry), medical and family history, and physical examination before inclusion. At baseline all subjects will be examined with single photon emission computed tomography (SPECT), MRI, fMRI, psychophysiology, neurocognition. In addition, they will be screened for drugs, genetic testing, and ECG. Patients will further be examined with clinical validated rating scales to measure psychopathology, subjective well-being, and side-effects. After a period of 6 weeks all assessments are repeated. During that period patients will be treated with amisulpride, while healthy controls will receive no treatment at all. Efficacy of antipsychotic treatment will be evaluated after this initial period of 6 weeks. Based on this evaluation it will be decided to either continue the current (amisulpride) antipsychotic treatment, or to switch to aripiprazole. Efficacy of aripiprazole is evaluated on a monthly basis, if the patient does not respond well enough, than the treatment will be adapted individually. Regardless of treatment, all subjects will be re-assessed in the same test battery as mentioned above, except for SPECT and fMRI, after a period of 6, 12, and 24 months. The developement in specific disturbances and the relationship between these will be analysed.

ELIGIBILITY:
Inclusion Criteria:

For patients: meeting diagnostic criteria for schizophrenia according to ICD 10 or DSM IV antipsychotic naive The controls will be matched to the patients according to gender age and parental socio-economic status.

-

Exclusion Criteria:

Patients: mental retardation, other chronic diseases, use of antidepressive medicine during the last month,being pregnant, on going substance abuse

Controls: psychiatric diagnosis, psychiatric diagnosis in first-degree relatives,on going drug abuse, mental retardation -

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2008-12; Primary Completion 2014-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Relationship between specific neuropsychiatric measures and improvement on PANSS scores | 6 weeks of medical treatment

SECONDARY OUTCOMES:
The relation between D2 binding potential (SPECT) and reward related brain activity (fMRI BOLD response) before and after D2 blockade | Baseline, 6 weeks
Time/dose improvement on PPI and other psychophysiological measures of early information processing after D2 blockade | Baseline, 2 and 6 weeks, 6,12,24 months
Disturbances in reward related fMRI BOLD response in antipsychotic naive schizophrenic patients | Baseline and 6 weeks follow up
Structural changes in grey and white matter before and after D2 blockade | 6 weeks, 6, 12 and 24 months,
Cognitive differences at baseline and changes over time after D2 blockade | Baseline, 6 weeks, 6,12,24 months
The effect of D2 blockade on reward related fMRI BOLD response | 6 weeks of medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Birte Y Glenthoj, professor, Study Director — University of Copenhagen, Psychiatric Center Glostrup, Ndr. Ringvej, DK-2600 Glostrup, Denmark
Locations (1):
- Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychiatric Center Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas MB, Raghava JM, Pantelis C, Rostrup E, Nielsen MO, Jensen MH, Glenthoj BY, Mandl RCW, Ebdrup BH, Fagerlund B. Associations between cognition and white matter microstructure in first-episode antipsychotic-naive patients with schizophrenia and healthy controls: A multivariate pattern analysis. Cortex. 2021 Jun;139:282-297. doi: 10.1016/j.cortex.2021.03.003. Epub 2021 Mar 18. PMID 33933719
- [Derived] Wulff S, Nielsen MO, Rostrup E, Svarer C, Jensen LT, Pinborg L, Glenthoj BY. The relation between dopamine D2 receptor blockade and the brain reward system: a longitudinal study of first-episode schizophrenia patients. Psychol Med. 2020 Jan;50(2):220-228. doi: 10.1017/S0033291718004099. Epub 2019 Jan 15. PMID 30642415
- [Derived] Ebdrup BH, Axelsen MC, Bak N, Fagerlund B, Oranje B, Raghava JM, Nielsen MO, Rostrup E, Hansen LK, Glenthoj BY. Accuracy of diagnostic classification algorithms using cognitive-, electrophysiological-, and neuroanatomical data in antipsychotic-naive schizophrenia patients. Psychol Med. 2019 Dec;49(16):2754-2763. doi: 10.1017/S0033291718003781. Epub 2018 Dec 18. PMID 30560750
- [Derived] Jessen K, Mandl RCW, Fagerlund B, Bojesen KB, Raghava JM, Obaid HG, Jensen MB, Johansen LB, Nielsen MO, Pantelis C, Rostrup E, Glenthoj BY, Ebdrup BH. Patterns of Cortical Structures and Cognition in Antipsychotic-Naive Patients With First-Episode Schizophrenia: A Partial Least Squares Correlation Analysis. Biol Psychiatry Cogn Neurosci Neuroimaging. 2019 May;4(5):444-453. doi: 10.1016/j.bpsc.2018.09.006. Epub 2018 Sep 25. PMID 30420252
- [Derived] Jessen K, Rostrup E, Mandl RCW, Nielsen MO, Bak N, Fagerlund B, Glenthoj BY, Ebdrup BH. Cortical structures and their clinical correlates in antipsychotic-naive schizophrenia patients before and after 6 weeks of dopamine D2/3 receptor antagonist treatment. Psychol Med. 2019 Apr;49(5):754-763. doi: 10.1017/S0033291718001198. Epub 2018 May 8. PMID 29734953
- [Derived] Anhoj S, Odegaard Nielsen M, Jensen MH, Ford K, Fagerlund B, Williamson P, Glenthoj B, Rostrup E. Alterations of Intrinsic Connectivity Networks in Antipsychotic-Naive First-Episode Schizophrenia. Schizophr Bull. 2018 Oct 17;44(6):1332-1340. doi: 10.1093/schbul/sbx171. PMID 29373756
- [Derived] Nielsen MO, Rostrup E, Wulff S, Bak N, Broberg BV, Lublin H, Kapur S, Glenthoj B. Improvement of brain reward abnormalities by antipsychotic monotherapy in schizophrenia. Arch Gen Psychiatry. 2012 Dec;69(12):1195-204. doi: 10.1001/archgenpsychiatry.2012.847. PMID 22868877
- See also: homepage of the research unit — http://www.cinsr.dk/
- See also: homepage of the research unit — http://www.cnsr.dk/